CLINICAL TRIAL: NCT04094597
Title: Effectivness and Safety of Oral Bovine Lactoferrin in Neonatal Sepsis and Necrotizing Enterocolitis and Its Effect on Anaemia of Prematurity
Brief Title: Safety and Efficacy of Oral Bovine Lactoferrin
Acronym: Lactoferrin
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, ayman zaher, Resident of Pediatrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Abu Elrich children hospital; 01525316 (Registry Identifier: Lactoferrin for prevention of neonatal sepsis)
Record Dates: First submitted 2019-04-04; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Neonatal SEPSIS
Keywords: lactoferrin
MeSH Terms: conditions — Neonatal Sepsis | interventions — Lactoferrin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: placebo group 100 patient will receive 2 ml saline for one month in comparison with oral lactoferrin for the same period to another 100 patient
Who Masked: Investigator
Masking Description: Follow up of the patients with CRP and different cultures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): saline is given orally in dose of 2 ml per day for one month
  Interventions: Drug: Placebos
- lacoferrin (Active Comparator): Pravotin is given orally 100 mg per sachet dissolved in 5 ml water given for one month
  Interventions: Drug: Lactoferrin

INTERVENTIONS:
Drug: Lactoferrin — lactoferrin is given orally in comparsion to placebp
  Other Names: Pravotin sachets
  Arms: lacoferrin
Drug: Placebos — placebp is given in 2 ml saline
  Other Names: saline
  Arms: placebo

SUMMARY:
Oral lactoferrin versus Placebo will be given to preterm neonates

DETAILED DESCRIPTION:
200 patient were included in the study , one hundred received oral placebo in the form of 2 ml saline , the other 100 preterm neonates received oral lactoferrin with monitoring of C-reactive protein , different cultures, complete blood count on day 7 and after one month.

ELIGIBILITY:
Inclusion Criteria:

All neonates born at Cairo university hospital NICU

Exclusion Criteria:

* Neonatal deaths before 3 days postnatal .
* Neonates with underlying gastrointestinal problems that prevent oral intake.
* Neonates with major congenital anomalies .
* Neonates with severe hypoxic ischemic encephaloapathy .
* Neonates whose parents refuse to participate.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
Change in mortality rate of neonatal sepsis in preterm neonate | one year
  Neonates will be assessed by C-reactive protein and different cultures to identify Neonatal sepsis
Number of Preterm Neonates who will have long term Complication after one month of regular use of Lactoferrin | one year
  Neonates will be assessed for long term complication as necrotizing enterocolitis , retinoapathy of prematurity and bronchopulmonary dysplasia

CONTACTS AND LOCATIONS:
Overall Officials: ayman zaher, bachelor, Principal Investigator — Cairo University
Locations (1):
- Ayman, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Yes
lactoferrin improves the mortality rate of neonatal sepsis
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: all the time
Access Criteria: lactoferrin

REFERENCES:
- See also: lactoferrin — http://www.ncbi.nlm.nih.gov/pubmed/?term=lacoferrin

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT04094597/SAP_000.pdf